CLINICAL TRIAL: NCT04199507
Title: Comparison of Postural Disorders and Physical Fitness Parameters, Family Anxiety Level and Quality of Life Between Individuals With Autism and Healthy Individuals Who Continue Physical Activity Program
Brief Title: Physical Fitness in Autism
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Kübra Şahan, Principal Investigator, Hacettepe University
Other Study IDs: GO18/905
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism: Assessment of physical activity level and physical fitness
  Interventions: Other: physical fitness assessment
- Healthy: Assessment of physical activity level and physical fitness
  Interventions: Other: physical fitness assessment

INTERVENTIONS:
Other: physical fitness assessment — assessment

SUMMARY:
Although there are some studies investigating the physical activity levels of children with autism in the literature, no comprehensive study investigating the relationship between posture and physical fitness parameters, family anxiety level and quality of life of individuals with autism who have continued physical activity program has not been found. The aim of our study is to compare postural disorders and physical fitness parameters, family anxiety level and quality of life between individuals with autism and healthy individuals attending physical activity program.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with mild to moderate autism,
2. To have the ability to emulate,
3. To have a cognitive level and cooperation capacity that will not hinder the implementation of assessment scales,

Exclusion Criteria:

1. Having any systemic chronic disease and neurological disorder
2. During the last 6 months, individuals wih autism in the process will affect physical fitness for fracture, surgery and so on.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Autism is a spectrum disorder, each person with autism has a distinct set of strengths and challenges. The ways in which people with autism learn, think and problem-solve can range from highly skilled to severely challenged. Some people with ASD may require significant support in their daily lives, while others may need less support and, in some cases, live entirely independently.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Physical fitness | 1 month
  Münich fitness test

SECONDARY OUTCOMES:
Posture analysis | 1 month
  New york posture analysis
Physical activity level | 1 month
  Godin leisure time activity questionnaire
Family Anxiety Level | 1 month
  State-Trait Anxiety Inventory: Scores range from 20 to 80. Scores are positively correlated with higher levels of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No